CLINICAL TRIAL: NCT03977961
Title: The Six-Minute Walking Test (6MWT) as a Measure of Functional Impairment in Lumbar Degenerate Disc Disease.
Acronym: 6MWT-DDD
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: PD Dr. med. Martin Stienen, Klinik für Neurochirurgie, Universitätsspital Zürich (Unknown); PD Dr. med. Oliver Gautschi, Neuro- und Wirbelsäulen Zentrum Zentral-schweiz, Luzern (Unknown)
Responsible Party: Principal Investigator, Nicolai Maldaner, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: 6MWT DDD - 1.0
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Disease; Lumbar Spine Degeneration; Lumbar Spinal Stenosis
MeSH Terms: conditions — Intervertebral disc disease; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DDD Patients: All patients presenting to the neurosurgical department of the Kantonsspital St. Gallen (KSSG) with a diagnosed DDD fulfilling the inclusion criteria and scheduled for surgery will be considered for this study.

SUMMARY:
The study determines the reliability and validity of the 6-Minute Walking Test (6MWT) in patients with lumbar degenerative disc disease (DDD).

DETAILED DESCRIPTION:
The purposes of the study is to assess the ability of the 6-Minute Walking Test (6MWT) as a reliable and standardized objective outcome assessment and its relation to already established subjective patient reported outcome measures in patients suffering from lumbar degenerative disc disease. We want to use an existing smartphone-application that uses global positioning system (GPS) coordinates to measure walking distance. Applying self- measurement of the 6MWT before and after a therapeutic intervention, we determine objective functional impairment (OFI) in patients. The results of this study add to the understanding of achievable objective outcomes after therapeutic interventions applied to patients with DDD and examines patients acceptance for smartphone based self-measurement.

Primary Objectives The primary objective is to determine the reliability and validity of the 6-Minute Walking Test (6MWT) in patients with lumbar degenerative disc disease (DDD)

Secondary objectives are

1. to correlate objective functional impairment (OFI) with already established patient-rated outcome measures (PROMs) in the sense of cross-validation.
2. To correlate OFI, as determined by the 6MWT with OFI that is determined by another objective test, the TUG test
3. to then analyze the change in OFI in patients before and after surgical intervention
4. to determine whether patients prefer the objective (6MWT) or subjective (PROMs) repeated assessment of their functional condition.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for spine surgery with one of the following diagnosis (1) lumbar disc herniation (LDH), (2) lumbar spinal stenosis lumbar (LSS) or lumbar DDD with or without instability requiring lumbar fusion (transforaminal lumbar interbody fusion, posterior lumbar interbody fusion, or extreme lateral interbody fusion)
* Male and Female subjects ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Inability to walk (extreme pain or severe neurological deficits)
* Severe Chronic Obstructive Lung Disease (COPD) corresponding to ≥ Gold III
* Severe heart failure corresponding to ≥ New York Heart Association (NYHA) III
* Lung cancer and diffuse parenchymal lung disease
* Other medical reasons interfering with the patient's ability to walk and perform the 6MWT (e.g., osteoarthritis disease of the lower extremities, Parkinson's disease, heart failure, hip or knee prosthesis etc.)
* Unavailability for follow up and/or inability to complete assessment (planning to move, no smartphone, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the neurosurgical department of the Kantonsspital St. Gallen (KSSG) with a diagnosed DDD fulfilling the inclusion criteria and scheduled for surgery will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Raw walking distance | 4-12 weeks
  Raw walking distance (in m), as measured with the 6MWT, between the baseline- (before surgery) and follow-up assessment

SECONDARY OUTCOMES:
TTFS | 4-12 weeks
  Difference in Time to First Symptoms (TTFS; in sec) as measured by the 6MWT, between the baseline- and follow-up assessment
DTFS | 4-12 weeks
  Difference in Distance to First Symptoms (DTFS, in m), as measured by the 6MWT, between the baseline- and follow-up assessment
Zurich Claudication Questionnaire (ZCQ) | 4-12 weeks
  Difference in PROM, as measured by the Zurich Claudication Questionnaire (ZCQ average score, range 0 (best) - 4,5 (worst), between the baseline- and follow-up assessment.
Core Outcome Measures Index (COMI) | 4-12 weeks
  Difference in health-related quality of life (hrQoL), as measured by the Core Outcome Measures Index (COMI average score, range 0 (best) - 10 (worst)), between the baseline- and follow-up assessment
TTFS/ZCQ baseline | 4-12 weeks
  Correlation of TTFS/DTFS in the 6MWT with the ZCQ score at baseline
TTFS/ZCQ follow-up | 4-12 weeks
  Correlation of TTFS in the 6MWT with the ZCQ score at follow-up
TTFS/COMI baseline | 4-12 weeks
  Correlation of TTFS/DTFS in the 6MWT with the COMI score at baseline
TTFS/COMI follow-up | 4-12 weeks
  Correlation of TTFS/DTFS in the 6MWT with the COMI score at follow-up
TTFS/TUG baseline | 4-12 weeks
  Correlation of TTFS/DTFS in the 6MWT with the Timed up go Test (TUG) at baseline
TTFS/TUG follow-up | 4-12 weeks
  Correlation of TTFS/DTFS in the 6MWT with the TUG at follow-up
Test-retest reliability of the 6MWT | 6 weeks to 1 day before surgery as well as 4-12 weeks after surgery
  Test-retest reliability of the 6MWT in patients with lumbar degenerate disc disease, tested two consecutive times with the 6MWT App (within 3 days) before as well as after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Maldaner, MD, Principal Investigator — Department of Neurosurgery
Locations (1):
- Kantonsspital St. Gallen / Department of Neurosurgery, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziga M, Sosnova M, Zeitlberger AM, Regli L, Bozinov O, Weyerbrock A, Ratliff JK, Stienen MN, Maldaner N. Objective outcome measures may demonstrate continued change in functional recovery in patients with ceiling effects of subjective patient-reported outcome measures after surgery for lumbar degenerative disorders. Spine J. 2023 Sep;23(9):1314-1322. doi: 10.1016/j.spinee.2023.05.002. Epub 2023 May 13. PMID 37182704
- [Derived] Zeitlberger AM, Sosnova M, Ziga M, Gautschi OP, Regli L, Bozinov O, Weyerbrock A, Stienen MN, Maldaner N. Distance to first symptoms measured by the 6-min walking test differentiates between treatment success and failure in patients with degenerative lumbar disorders. Eur Spine J. 2022 Mar;31(3):596-603. doi: 10.1007/s00586-021-07103-9. Epub 2022 Jan 11. PMID 35015137
- [Derived] Zeitlberger AM, Sosnova M, Ziga M, Regli L, Bozinov O, Weyerbrock A, Stienen MN, Maldaner N. Assessment of the Minimum Clinically Important Difference in the Smartphone-based 6-minute Walking Test After Surgery for Lumbar Degenerative Disc Disease. Spine (Phila Pa 1976). 2021 Sep 15;46(18):E959-E965. doi: 10.1097/BRS.0000000000003991. PMID 34042414
- [Derived] Maldaner N, Sosnova M, Ziga M, Zeitlberger AM, Bozinov O, Gautschi OP, Weyerbrock A, Regli L, Stienen MN. External Validation of the Minimum Clinically Important Difference in the Timed-up-and-go Test After Surgery for Lumbar Degenerative Disc Disease. Spine (Phila Pa 1976). 2022 Feb 15;47(4):337-342. doi: 10.1097/BRS.0000000000004128. PMID 34033596
- [Derived] Maldaner N, Sosnova M, Zeitlberger AM, Ziga M, Gautschi OP, Regli L, Bozinov O, Weyerbrock A, Stienen MN. Responsiveness of the self-measured 6-minute walking test and the Timed Up and Go test in patients with degenerative lumbar disorders. J Neurosurg Spine. 2021 May 7;35(1):52-59. doi: 10.3171/2020.11.SPINE201621. Epub 2021 May 7. PMID 33974372